CLINICAL TRIAL: NCT02225457
Title: Study of the Determinants and Mechanisms of Adaptation of Metabolic Responses to Controlled Overfeeding in Female and Male Healthy Volunteers
Brief Title: Study of the Mechanisms of Metabolic Adaptations to Overfeeding
Acronym: Polynut
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: University of Lyon (Other)
Responsible Party: Principal Investigator, Francois Pralong, Full Professor and Head, Cervice of Endocrinology, Diabetology and Metabolism, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 391/13; SNF 320030_141065 (Other Grant/Funding Number: Swiss National Science Foundation)
Record Dates: First submitted 2014-07-21; First posted 2014-08-26 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Obesity; Diabetes
Keywords: insulin resistance; type 2 diabetes; obesity; polyphenols; adipose tissue; overfeeding
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Insulin Resistance; Diabetes Mellitus, Type 2 | interventions — Polyphenols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypercaloric diet and polyphenols (Experimental): polyphenols will consist in the administration of 1 gram (5x200 mg) of the compound bid during the entire overfeeding period.
  Hypercaloric diet will consist in a hypercaloric diet providing an excess of 50% KCal over daily requirements, and will last 30 days.
  Interventions: Other: Hypercaloric diet; Dietary Supplement: polyphenols
- Hypercaloric diet and placebo (Active Comparator): Placebo will consist in the administration of a number of placebo pills matching that of polyphenols, in a similar way (bid) for the duration of the overfeeding experiment.
  Overfeeding will consist in a hypercaloric diet providing an excess of 50% KCal over daily requirements, and will last 30 days.
  Interventions: Other: Hypercaloric diet; Dietary Supplement: placebo (for polyphenols)

INTERVENTIONS:
Other: Hypercaloric diet — Hypercaloric diet will be designed to provide 50% excess in calories compared to daily requirements. It will consist in a "snack" type, high fat and high carbohydrates diet.
  Other Names: Overfeeding
Dietary Supplement: polyphenols — Administration of polyphenols will consist in the administration of 1 gram (5x200 mg) of the compound bid during the entire overfeeding period.
  Arms: Hypercaloric diet and polyphenols
Dietary Supplement: placebo (for polyphenols) — Placebo will consist in the administration of a number of placebo pills matching that of polyphenols, in a similar way (bid) for the duration of the overfeeding experiment.
  Arms: Hypercaloric diet and placebo

SUMMARY:
Obesity results from complex interactions between genetic and environmental factors, and are strongly associated with metabolic complications such as type 2 diabetes mellitus. Obesity is defined as an excessive fat accumulation that presents a risk to health, a risk that is highly dependent upon the type of adipose tissue accumulation, whether visceral or sub-cutaneous, but also upon the characteristics of the fat tissue, especially inflammatory cells accumulation. Because of the well known sexual difference in fat accretion, this obesity-associated risk may also be very different for men and for women. In addition, recent data indicate that various factors such as the intestinal microbiota, but also the dietary intake of protective nutrients might be important determinants of the metabolic complications of obesity.

Here we propose to: 1) study the metabolic adaptations and the mechanisms of adipose tissue accumulation during a period of controlled caloric over-nutrition, both in men and in women; 2) evaluate the potential protective effects of a supplementation with polyphenols on insulin resistance and other metabolic adaptations.

DETAILED DESCRIPTION:
To achieve these goals, healthy male and female volunteers will be enrolled into a one month longitudinal, prospective study on the influence of hypercaloric overfeeding (+50% of daily caloric needs) on different tissues (adipose tissue, muscle and blood).

They will be separated into two different groups: hypercaloric nutrition and placebo, and hypercaloric nutrition and polyphenols (2g/day), where polyphenols administration will be randomized and administered in a double blind fashion. Whole body and hepatic insulin sensitivity, total energy expenditure, glucose hepatic production, protein and gene expression in muscle, adipose tissue and blood as well as intestinal microbiota will be assessed at base line, and after one month of overfeeding.

ELIGIBILITY:
Inclusion Criteria:

* normal healthy male and female volunteer

Exclusion Criteria:

* Diabetes mellitus
* High blood pressure
* Liver disease
* Kidney disease

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-05 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in insulin sensitivity | baseline, day 31 of overfeeding
  Whole body insulin sensitivity will be measured during hyperinsulinemic, euglycemic clamps.

SECONDARY OUTCOMES:
Change from baseline in muscle and adipose tissue gene expression | Baseline, day 28 of overfeeding
  Transcriptomic experiments will be performed on muscle and adipose tissue samples

CONTACTS AND LOCATIONS:
Overall Officials: Francois P Pralong, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- CHUVaudois, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Bartova S, Madrid-Gambin F, Fernandez L, Carayol J, Meugnier E, Segrestin B, Delage P, Vionnet N, Boizot A, Laville M, Vidal H, Marco S, Hager J, Moco S. Grape polyphenols decrease circulating branched chain amino acids in overfed adults. Front Nutr. 2022 Oct 26;9:998044. doi: 10.3389/fnut.2022.998044. eCollection 2022. PMID 36386937
- [Derived] Segrestin B, Delage P, Nemeth A, Seyssel K, Disse E, Nazare JA, Lambert-Porcheron S, Meiller L, Sauvinet V, Chanon S, Simon C, Ratiney H, Beuf O, Pralong F, Yassin NA, Boizot A, Gachet M, Burton-Pimentel KJ, Vidal H, Meugnier E, Vionnet N, Laville M. Polyphenol Supplementation Did Not Affect Insulin Sensitivity and Fat Deposition During One-Month Overfeeding in Randomized Placebo-Controlled Trials in Men and in Women. Front Nutr. 2022 May 9;9:854255. doi: 10.3389/fnut.2022.854255. eCollection 2022. PMID 35614978